CLINICAL TRIAL: NCT04139629
Title: Cohort Study Investigating the Association Between Antichlamydial Antibody Positivity and Efficiency of Treatment With Assisted Reproduction Technologies (ART) in Women With Tubal Factor Infertility
Brief Title: Cohort Study Investigating the Association Between Antichlamydial Antibody Positivity and ART Outcomes in Women With TFI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: D.O. Ott Research Institute of Obstetrics, Gynecology, and Reproductology (Other)
Responsible Party: Principal Investigator, Valeria Muller, Doctor at IVF department, D.O. Ott Research Institute of Obstetrics, Gynecology, and Reproductology
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: D-19
Record Dates: First submitted 2019-10-21; First posted 2019-10-25 (Actual); Last update posted 2021-08-24 (Actual); Status verified 2021-08

CONDITIONS: Antichlamydial Antibodies; Chlamydia Trachomatis Infection; Infertility; Tubal Factor Infertility
Keywords: Antichlamydial antibodies; in vitro fertilization; ovarian stimulation; tubal factor infertility
MeSH Terms: conditions — Infertility | interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- antibody positive (CAT+) (Other): patients found positive for one of the assayed antichlamydial antibodies
  Interventions: Diagnostic Test: antichlamydial antibody test; Drug: treatment of infertility with ART
- antibody negative (CAT-) (Other): women with negative antichlamydia antibody test
  Interventions: Diagnostic Test: antichlamydial antibody test; Drug: treatment of infertility with ART

INTERVENTIONS:
Diagnostic Test: antichlamydial antibody test — At the first day of stimulation blood analyses for IgG, IgA and IgM (ELISA) to major chlamydial antigens (anti-C.trachomatis), major outer membrane protein (MOMP) and plasmid-encoded protein (pgp3) will be performed for patients found eligible for the study.
Drug: treatment of infertility with ART — COS in gonadotropin-releasing hormone (GnRH) antagonist protocol with IVF/ICSI, fresh ET and, if no pregnancy occurred, frozen/thawed ET (for all embryos resulting from this COS) will be performed.
  Other Names: Procedure

SUMMARY:
In a prospective cohort study investigators will examine characteristics and clinical outcomes of treatment with ART in women with tubal factor infertility (TFI) with regard to seropositivity to antichlamydial antibodies.

DETAILED DESCRIPTION:
At the first day of stimulation blood analyses for immunoglobulin G (IgG), immunoglobulin A (IgA) and immunoglobulin M (IgM) to major chlamydial antigens (anti-C.trachomatis), major outer membrane protein (MOMP) and plasmid-encoded protein (pgp3) will be performed for patients found eligible for the study.

According to the result of chlamydial antibody test (CAT) participants will be divided into two groups: group A - women with at least one of antibodies detected (CAT+); Group B - seronegative subjects (CAT-).

Women of both groups will undergo a conventional ovarian stimulation (COS) with GnRH antagonist and daily gonadotropin administration at the dose of 150-300 international unit (IU).

Retrieved oocytes following fertilization (conventional IVF or ICSI) will be cultured to Day 3-5 in vitro; ultrasound guided single or double embryo transfer will be performed; remaining embryos of eligible quality will be vitrified.

Patients will be followed up to live birth. Frozen/thawed embryo transfers (FET) will be performed until at least one live birth (≥20 weeks of gestation) occurred or all embryos resulting from the mentioned assisted ovarian stimulation were used.

ELIGIBILITY:
Inclusion Criteria:

* Tubal factor infertility diagnosed by laparoscopy;
* Female age between 20-41 years;
* BMI 17,5-35 kg/m2;
* Early follicular phase follicle stimulating hormone (FSH) ≤15 IU/L
* Presence of viable spermatozoa in partner's sperm;
* Signed informed consent.

Exclusion Criteria:

* previous ovarian surgery;
* endometriosis;
* antimullerian hormone (AMH) level ≤0,3 ng/ml;
* hyper- or hypogonadotropic ovarian failure;
* severe male factor infertility;
* Pre-existing medical condition preventing or interfering with IVF treatment: any clinically significant systemic disease; inherited or acquires thrombophilia and thromboembolism; endocrine or metabolic abnormalities; moderate or severe impairment of renal or hepatic function; any oncological diseases in anamnesis; known history of recurrent miscarriage, abnormal karyotype of both partners; currently active pelvic inflammatory disease;
* Abnormal IVF screening tests: Papanicolaou (PAP) smear, Syphilis, HIV 1&2, Hepatitis B, Hepatitis C, Chlamydia, and Gonorrhea;
* Presence of uterine pathology: Asherman's Syndrome, endometrial polyps, nodus form of adenomyosis or uterine fibroids ≥3 mm in diameter;
* Visualization of ovarian cysts ≥25 mm, endometriomas or hydrosalpinx;
* One or more follicles ≥8 mm at the start of the COS protocol.

Ages: 20 Years to 41 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 292 (Actual)
Dates: Start 2019-10-25 (Actual); Primary Completion 2020-01-30 (Actual); Study Completion 2021-10-30 (Estimated)

PRIMARY OUTCOMES:
number of oocytes (COCs) | 2-4 weeks after after assignment (at oocyte recovery day)
  obtained during oocyte pick-up (OPU)

SECONDARY OUTCOMES:
Number of low prognostic patients | up to 1 week after assignment
  according to POSEIDON criteria low prognostic patients will be divided to 4 groups
Duration of stimulation | 2-4 weeks after assignment
  total days of COS: from the first gonadotropins administration to ovulation triggering
Number/rate of participants with poor or suboptimal response to COS | 2-4 weeks after after assignment (at oocyte recovery day)
  ≤5, 5-9 cumulus-oocyte complexes (COCs) at OPU respectively
Number / rate of mature (MII) oocytes | 2-4 weeks after after assignment (at oocyte recovery day)
  assessment is done only for ICSI cycles
Fertilization rate | at day 1 after oocyte recovery
  number / rate of two-pronuclear zygotes (2PN) on day 1 after fertilization
Number / rate of best and good quality embryos per transfer | 3-5 weeks after after assignment (at ET day)
  embryo quality assessment according to known classifications
Implantation rate | 3-4 weeks after fresh or frozen/thawed ET
  ratio of the number of intrauterine gestational sac (at 5-6 weeks of gestation) to the number of transferred embryos
clinical pregnancy rate | 5-6 weeks after starting the stimulation or 3-4 weeks after frozen/thawed ET
  presence of intrauterine gestational sac at transvaginal ultrasound at 5-6 weeks of gestation or 5-6 weeks after starting the intervention; measured per embryo transfer

OTHER OUTCOMES:
Live birth rate | up to 3 years after assignment
  at least one live born baby at ≥20 weeks of gestation; measured per oocyte aspiration, fresh embryo transfer
Cumulative live birth rate | up to 3 years after assignment
  at least one live born baby at ≥20 weeks of gestation from ART aspiration cycle, including fresh and frozen/thawed ET, resulting from assisted ovarian stimulation until one live birth occurred or all embryos were used
Cost-effectiveness of COS | up to 3 years after assignment
  ratio of total cost of stimulation, FETs to the number of patients with clinical pregnancy
Cycle cancellation rate | up to 2 years after assignment
  during COS (no response), at OPU (premature ovulation, absence or degradation of COCs), during in vitro cultivation and thawing (fertilization failure, inadequate embryo quality), other reasons (adverse events, hyper stimulation syndrome, withdrawal);

CONTACTS AND LOCATIONS:
Overall Officials: Alexandr Gzgzyan, Prof, PhD, Principal Investigator — D.O. Ott Research Institute of Obstetrics, Gynecology, and Reproductology
Locations (1):
- D.O. Ott Research Institute of Obstetrics, Gynecology and Reproductology, Saint Petersburg, Russia

IPD SHARING:
Plan to Share IPD: Yes
at the end of recruitment ICF and brief CRF will be shared. At the study completion - CSR and SAP will be uploaded
Supporting Information: SAP, ICF, CSR
Time Frame: at the study completion for 1 year
Access Criteria: 30 random CRFs will be shared, more by request